CLINICAL TRIAL: NCT00002099
Title: Phase II/III Study of the Tolerance and Efficacy of Combined Use of Didanosine (2',3'-Dideoxyinosine; ddI) and Lentinan in HIV-Positive Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AJI Pharma USA (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 126B; 92-11-9
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-07

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Lentinan
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Lentinan; Didanosine

INTERVENTIONS:
Drug: Lentinan
Drug: Didanosine

SUMMARY:
To determine the tolerance and side effects of a combination of lentinan and didanosine (ddI) in comparison with ddI alone. To determine whether the combination of lentinan and ddI produces a significant immunorestorative effect within the study observation period (6-12 months) as measured by an increase in one or more of the following: neutrophil count and activity, T-cell subsets, and a decrease in p24 antigen.

DETAILED DESCRIPTION:
Patients are treated with daily oral ddI for 6 weeks, then are randomized to ddI in combination with intravenous lentinan or placebo (administered once weekly) for 26 weeks. Patients who are already stabilized on 400 mg/day ddI will proceed directly to randomization. Following completion of the combination therapy, patients may be offered 26 additional weeks of therapy on an optional basis.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity.
* Absolute CD4 count of 200 - 500 cells/mm3.
* No active opportunistic infection or Kaposi's sarcoma.

Prior Medication:

Allowed:

* Prior ddI for no longer than 3 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Lymphoid malignancy.
* Pancreatitis.
* Peripheral neuropathy.
* Critical illness.

Concurrent Medication:

Excluded:

* Antiretroviral agents other than ddI.
* Steroids.
* Cytotoxic agents.
* Immunosuppressive agents.
* Immunomodulators.
* 1-Thyroxine.

Concurrent Treatment:

Excluded:

* Radiotherapy.

Prior Medication:

Excluded within 1 month prior to study entry:

* Antiretroviral agents other than ddI (patients may have received prior ddI for no longer than 3 months total).
* Steroids.
* Cytotoxic agents.
* Immunosuppressive agents.
* Immunomodulators.

Prior Treatment:

Excluded:

* Radiotherapy within 1 month prior to study entry. Active IV drug abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pearce D, Study Chair
Locations (1):
- HIV Research Group, San Diego, California, United States